CLINICAL TRIAL: NCT00271050
Title: The Role of Conformal External Beam Radiotherapy in the Management of Patients With Bulky Disease Undergoing Y90-Ibritumomab Tiuxetan (Zevalin) Radio-immunotherapy for Indolent B-cell Non-Hodgkin's Lymphoma
Brief Title: External Beam Radiotherapy and Zevalin for Management of Indolent B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Roger Macklis, MD, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 7883; CCF IRB 7883; Case 1405
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Lymphoma, B-Cell
Keywords: non-Hodgkin's lymphoma; external beam radiotherapy (EBRT); radio-immunotherapy (RIT); Zevalin
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

ARMS (1):
- 1 (Experimental)
  Interventions: Other: external beam radiotherapy plus 90-Y ibritumomab tiuxetan

INTERVENTIONS:
Other: external beam radiotherapy plus 90-Y ibritumomab tiuxetan — combination of EBRT followed by radioimmunotherapeutic 90-Y ibritumomab tiuxetan
  Other Names: Zevalin

SUMMARY:
The purpose of the research study is to learn whether external beam radiation can be used as a safe and effective treatment for patients with bulky (≥ 5cm) sites of non-Hodgkin's lymphoma prior to treatment with 90Y-ibritumomab tiuxetan (Zevalin).

DETAILED DESCRIPTION:
Non-Hodgkin's lymphomas (NHL) are a heterogeneous group of lymphoid malignancies that represent the 6th leading cause of cancer death and the 2nd fastest growing cancer in the United States. NHLs can be divided into two prognostic groups: aggressive and indolent lymphomas. Aggressive NHLs grow rapidly and present as disseminated disease in 70% of cases, yet can be cured in a significant number of patients with intensive combination chemotherapy regimens. Indolent (low-grade) NHLs are slow growing malignancies with long natural histories that are incurable when disseminated. Early stage low-grade NHL (stage I and II) has the potential for cure with radiotherapy, but only 10-20% of patients with low-grade NHL present with early stage disease. The vast majority of patients with low-grade NHL present with advanced disseminated disease. While indolent B-cell NHLs have initial sensitivity to chemotherapy and radiotherapy, they frequently relapse and become increasingly resistant to therapy with each successive relapse, eventually transforming to aggressive lymphomas in most patients. Fifty percent of patients presenting with advanced indolent NHL die within 5 years of their first relapse. Only modest improvement has been made in the last 25 years in increasing the survival of patients with indolent NHL with current median survival of 7-10 years.

Recent advances in the field of immunotherapy have proved to benefit patients with relapsed or refractory B-cell NHL. In 1997, rituximab became the first FDA-approved monoclonal antibody (mAb) for the treatment of cancer. Rituximab, a chimeric IgG1 kappa monoclonal antibody, specifically recognizes and binds to the CD20 antigen found on the cell surface of most normal B-cells and malignant B-cell lymphomas. Rituximab binds human complement and lyses B-cell lines through complement dependent cytotoxicity and antibody dependent cellular toxicity. A multi-center Phase II trial of 166 patients with relapsed indolent B-cell lymphoma treated with rituximab found an overall response in 50% of patients with 6% having a complete response and 44% having a partial response. Time to progression was a median of 13 months in patients who responded.

The introduction of radioimmunotherapy (RIT) has exploited the tumor cell targeting ability of mAbs to deliver doses of radiation to the tumor and limited surrounding tissue. This is especially useful in the treatment of NHL because lymphomas are highly sensitive to radiotherapy. 90Yttrium-ibritumomab tiuxetan (Zevalin) is a unique compound composed of the murine IgG1 anti-CD20 antibody ibritumomab, the linker chelator tiuxetan, and the radioisotope 90Y chelated via the linker. 90Y-ibritumomab tiuxetan can be described as providing a double hit therapeutic approach by having the CD20+ antibody properties of rituximab combined with radiation therapy.

90Yttrium-ibritumomab tiuxetan appears to be effective in the treatment of patients refractory to treatment with rituximab, but response rates decrease with increasing tumor size. 90Y-ibritumomab tiuxetan was approved by the FDA in 2002 for the treatment of patients with relapsed or refractory low-grade, follicular, or CD20+ transformed B-cell non-Hodgkin's lymphoma (NHL), and rituximab-refractory follicular NHL.

A preliminary survey of 20 patients treated with 90Y-ibritumomab tiuxetan at the Cleveland Clinic Foundation from 1998-2003 detailed patterns of NHL recurrence after treatment. The results of this survey were presented in part by Dr. Macklis at the 2004 annual meeting of the American Society of Therapeutic Radiation Oncology (ASTRO) in Atlanta and recently accepted for publication in the International Journal of Radiation Oncology, Biology, Physics. Based on preliminary data, a hypothesis can be made that some likely sites of disease recurrence/progression after RIT can be predicted by the volume of disease at a specific site prior to RIT. In short, pre-RIT bulky sites of disease are the most likely locations of disease recurrence after RIT followed by gross, but non-bulky, pre-RIT sites followed by entirely new sites. Based on this hypothesis, it might be beneficial to pre-treat bulky sites of NHL with external beam radiotherapy prior to RIT in order to promote a more durable response. Doses of external beam radiation required to consolidate these bulky disease sites are unclear.

In this study, we plan to utilize a dose of EBRT of 2,400cGy to bulky sites of disease followed by RIT. Though the combined effects of 2,400cGy of EBRT and RIT are likely to be well tolerated, such a combination has not been sufficiently studied. Therefore, the primary goal of this study is to determine if the combination of EBRT and RIT has an acceptable toxicity profile with regard to long-term myelosuppression and other non-hematological toxicities.

ELIGIBILITY:
Inclusion Criteria:

* B-cell non-Hodgkin's lymphoma of one of the following types as defined by the WHO classification:
* Small lymphocytic lymphoma/Chronic lymphocytic leukemia
* Nodal marginal zone B-cell lymphoma
* Extranodal marginal zone B-cell lymphoma
* Splenic marginal zone lymphoma
* Lymphoplasmacytic lymphoma
* Follicular lymphoma
* Diffuse large B-cell lymphoma which has transformed from one of the previously listed types of lymphomas
* At least one site of lymphoma greater than or equal to 5 cm in any dimension
* Received at least one prior therapy
* Should show evidence of symptomatology as a result of their disease and/or evidence of progression of their disease.
* Measurable disease using Cheson criteria [23] for Non-Hodgkin's Lymphoma: a lymph node that is greater than 1 cm in its longest transverse diameter by CT scan should be considered compatible with involvement by NHL
* No anti-cancer therapy for four weeks (six weeks if rituximab, nitrosourea or Mitomycin C) prior to study initiation, and fully recovered from all toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy
* An IRB-approved signed informed consent
* Age greater than or equal to 18
* Expected survival greater than or equal to 3 months
* Prestudy performance status of 0, 1, or 2 according to WHO
* Absolute neutrophil count ([segmented neutrophils + bands] x total WBC) > 1500/mm3 within two weeks prior to first dose of external beam radiation and also documented again two weeks prior to 90Y-ibritumomab tiuxetan treatment
* Platelet counts greater than or equal to 100,000 within two weeks prior to first dose of external beam radiation and also documented again two weeks prior to 90Y-ibritumomab tiuxetan treatment
* Bone marrow involvement by NHL less than 26% within six weeks of treatment with 90Y-ibritumomab tiuxetan
* Cellularity of bone marrow > 15% within 6 weeks of study
* Female patients who are not pregnant or lactating
* Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician, abstinence is an acceptable method)

Exclusion Criteria:

* Prior radioimmunotherapy
* Presence of CNS lymphoma
* Absolute lymphocyte count ≥ 5000
* HIV or AIDS-related lymphoma
* Large pleural effusions or ascites
* Total bilirubin > 2.0 mg/dL
* Serum creatinine > 2.0 mg/dL
* Patients who, in the opinion of their oncology team, have prior external beam radiation therapy to > 25% of active skeletal marrow (either involved field or regional)
* Patients who have received G-CSF or GM-CSF therapy within two weeks or pegfilgrastim within 4 weeks prior to treatment
* Serious nonmalignant disease or infection which, in the opinion of the investigator, would compromise other protocol objectives
* Major surgery, other than diagnostic surgery, within four weeks
* Pregnant women or women of child-bearing age who refuse pregnancy tests
* Patients who have had prior myeloablative autologous or allogenic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PET and CT (w/oral and IV contrast) | 90 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roger Macklis, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Fisher RI. Overview of non-Hodgkin's lymphoma: biology, staging, and treatment. Semin Oncol. 2003 Apr;30(2 Suppl 4):3-9. doi: 10.1053/sonc.2003.23797. PMID 12728402
- [Background] Dillman RO. Radiolabeled anti-CD20 monoclonal antibodies for the treatment of B-cell lymphoma. J Clin Oncol. 2002 Aug 15;20(16):3545-57. doi: 10.1200/JCO.2002.02.126. No abstract available. PMID 12177115
- [Background] Gustavsson A, Osterman B, Cavallin-Stahl E. A systematic overview of radiation therapy effects in non-Hodgkin's lymphoma. Acta Oncol. 2003;42(5-6):605-19. doi: 10.1080/02841860310014435. PMID 14596518
- [Background] Tobinai K. Rituximab and other emerging antibodies as molecular target-based therapy of lymphoma. Int J Clin Oncol. 2003 Aug;8(4):212-23. doi: 10.1007/s10147-003-0295-y. PMID 12955576
- [Background] Seymour JF. New treatment approaches to indolent non-Hodgkin's lymphoma. Semin Oncol. 2004 Feb;31(1 Suppl 2):27-32. PMID 15042532
- [Background] Forero A, Lobuglio AF. History of antibody therapy for non-Hodgkin's lymphoma. Semin Oncol. 2003 Dec;30(6 Suppl 17):1-5. doi: 10.1053/j.seminoncol.2003.10.002. PMID 14710396
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- [Background] Cheson BD. Radioimmunotherapy of non-Hodgkin lymphomas. Blood. 2003 Jan 15;101(2):391-8. doi: 10.1182/blood-2002-06-1793. Epub 2002 Sep 19. PMID 12393555
- [Background] Witzig TE, White CA, Wiseman GA, Gordon LI, Emmanouilides C, Raubitschek A, Janakiraman N, Gutheil J, Schilder RJ, Spies S, Silverman DH, Parker E, Grillo-Lopez AJ. Phase I/II trial of IDEC-Y2B8 radioimmunotherapy for treatment of relapsed or refractory CD20(+) B-cell non-Hodgkin's lymphoma. J Clin Oncol. 1999 Dec;17(12):3793-803. doi: 10.1200/JCO.1999.17.12.3793. PMID 10577851
- [Background] Witzig TE, Gordon LI, Cabanillas F, Czuczman MS, Emmanouilides C, Joyce R, Pohlman BL, Bartlett NL, Wiseman GA, Padre N, Grillo-Lopez AJ, Multani P, White CA. Randomized controlled trial of yttrium-90-labeled ibritumomab tiuxetan radioimmunotherapy versus rituximab immunotherapy for patients with relapsed or refractory low-grade, follicular, or transformed B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2002 May 15;20(10):2453-63. doi: 10.1200/JCO.2002.11.076. PMID 12011122
- [Background] Justice TE, Martenson JA, Wiseman GA, Witzig TE. External beam radiation therapy after 90Y-ibritumomab tiuxetan radioimmunotherapy for relapsed or refractory CD20+ non-Hodgkin's lymphoma. Int J Radiat Oncol Biol Phys 2003; 57(Suppl 2):S287-8
- [Background] O'Doherty MJ, Hoskin PJ. Positron emission tomography in the management of lymphomas: a summary. Eur J Nucl Med Mol Imaging. 2003 Jun;30 Suppl 1:S128-30. doi: 10.1007/s00259-003-1170-9. Epub 2003 Apr 12. No abstract available. PMID 12692689
- [Background] Blum RH, Seymour JF, Wirth A, MacManus M, Hicks RJ. Frequent impact of [18F]fluorodeoxyglucose positron emission tomography on the staging and management of patients with indolent non-Hodgkin's lymphoma. Clin Lymphoma. 2003 Jun;4(1):43-9. doi: 10.3816/clm.2003.n.013. PMID 12837154
- [Background] Kostakoglu L, Goldsmith SJ. Fluorine-18 fluorodeoxyglucose positron emission tomography in the staging and follow-up of lymphoma: is it time to shift gears? Eur J Nucl Med. 2000 Oct;27(10):1564-78. doi: 10.1007/s002590000340. PMID 11083548
- [Background] Leskinen-Kallio S, Ruotsalainen U, Nagren K, Teras M, Joensuu H. Uptake of carbon-11-methionine and fluorodeoxyglucose in non-Hodgkin's lymphoma: a PET study. J Nucl Med. 1991 Jun;32(6):1211-8. PMID 2045935
- [Background] Okada J, Yoshikawa K, Imazeki K, Minoshima S, Uno K, Itami J, Kuyama J, Maruno H, Arimizu N. The use of FDG-PET in the detection and management of malignant lymphoma: correlation of uptake with prognosis. J Nucl Med. 1991 Apr;32(4):686-91. PMID 2013808
- [Background] Newman JS, Francis IR, Kaminski MS, Wahl RL. Imaging of lymphoma with PET with 2-[F-18]-fluoro-2-deoxy-D-glucose: correlation with CT. Radiology. 1994 Jan;190(1):111-6. doi: 10.1148/radiology.190.1.8259386.
- [Background] Torizuka T, Zasadny KR, Kison PV, Rommelfanger SG, Kaminski MS, Wahl RL. Metabolic response of non-Hodgkin's lymphoma to 131I-anti-B1 radioimmunotherapy: evaluation with FDG PET. J Nucl Med. 2000 Jun;41(6):999-1005. PMID 10855624
- [Background] Scheidhauer K, Wolf I, Baumgartl HJ, Von Schilling C, Schmidt B, Reidel G, Peschel C, Schwaiger M. Biodistribution and kinetics of (131)I-labelled anti-CD20 MAB IDEC-C2B8 (rituximab) in relapsed non-Hodgkin's lymphoma. Eur J Nucl Med Mol Imaging. 2002 Oct;29(10):1276-82. doi: 10.1007/s00259-002-0820-7. Epub 2002 Jul 6. PMID 12271407
- [Background] Hofmann M, Hertenstein B, Boerner AR, Heil G, Peest D, Knoop BO, Geworski L, Otto D, Ganser A, Knapp WH. 18-F-FDG-PET in monitoring therapy response to RIT by 131-I Rituximab (Mabthera) antibody. Annals Onc 2002; 13 (Suppl 2): 96.
- [Background] Macklis R, Molina A, Pohlman B, Gordon L, Wang H, Saville MW, Witzig T. Long-term responses in patients with relapsed or refractory follicular lymphoma treated with yttrium 90 ibritumomab tiuxetan (Zevalin). Int J Radiat Oncol Biol Phys 2004; 60 (Suppl 1): S542 (2346).
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- [Background] Gordon LI, Molina A, Witzig T, Emmanouilides C, Raubtischek A, Darif M, Schilder RJ, Wiseman G, White CA. Durable responses after ibritumomab tiuxetan radioimmunotherapy for CD20+ B-cell lymphoma: long-term follow-up of a phase 1/2 study. Blood. 2004 Jun 15;103(12):4429-31. doi: 10.1182/blood-2003-11-3883. Epub 2004 Mar 11. PMID 15016644
- [Background] Witzig TE, White CA, Gordon LI, Wiseman GA, Emmanouilides C, Murray JL, Lister J, Multani PS. Safety of yttrium-90 ibritumomab tiuxetan radioimmunotherapy for relapsed low-grade, follicular, or transformed non-hodgkin's lymphoma. J Clin Oncol. 2003 Apr 1;21(7):1263-70. doi: 10.1200/JCO.2003.08.043. PMID 12663713
- [Background] Chen EX, Tannock IF. Risks and benefits of phase 1 clinical trials evaluating new anticancer agents: a case for more innovation. JAMA. 2004 Nov 3;292(17):2150-1. doi: 10.1001/jama.292.17.2150. No abstract available. PMID 15523076
- [Background] Eisenhauer EA, O'Dwyer PJ, Christian M, Humphrey JS. Phase I clinical trial design in cancer drug development. J Clin Oncol. 2000 Feb;18(3):684-92. doi: 10.1200/JCO.2000.18.3.684. PMID 10653884
- [Background] Yahalom J, Mauch P. The involved field is back: issues in delineating the radiation field in Hodgkin's disease. Ann Oncol. 2002;13 Suppl 1:79-83. doi: 10.1093/annonc/13.s1.79. PMID 12078908
- [Background] Josting A, Rudolph C, Mapara M, Glossmann JP, Sieniawski M, Sieber M, Kirchner HH, Dorken B, Hossfeld DK, Kisro J, Metzner B, Berdel WE, Diehl V, Engert A. Cologne high-dose sequential chemotherapy in relapsed and refractory Hodgkin lymphoma: results of a large multicenter study of the German Hodgkin Lymphoma Study Group (GHSG). Ann Oncol. 2005 Jan;16(1):116-23. doi: 10.1093/annonc/mdi003. PMID 15598948
- [Background] Chen Q, Chai YC, Mazumder S, Jiang C, Macklis RM, Chisolm GM, Almasan A. The late increase in intracellular free radical oxygen species during apoptosis is associated with cytochrome c release, caspase activation, and mitochondrial dysfunction. Cell Death Differ. 2003 Mar;10(3):323-34. doi: 10.1038/sj.cdd.4401148. PMID 12700632
- [Background] Kaminski MS, Leonard JP, Zelenetz AD, Vose JM. Bexxar therapy (tositumomab and iodine I-131) has high response rates in the treatment of bulky low grade relapsed or refractory non-Hodgkin's lymphoma. 2002 ASCO Annual Meeting. Abstract #17.